CLINICAL TRIAL: NCT04829721
Title: Pelvic Floor Disorder Assessment of Knowledge and Symptoms: an Educational Model in Spanish-Speaking Women
Acronym: PAKS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00236091
Record Dates: First submitted 2021-03-31; First posted 2021-04-02 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Pelvic Organ Prolapse; Urinary Incontinence; Patient Education
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational Video Workshop (Experimental): A single 20 minute video workshop on pelvic floor disorders.
  Interventions: Other: Educational Intervention with video

INTERVENTIONS:
Other: Educational Intervention with video — Women randomized to an educational video workshop group.

SUMMARY:
Pelvic floor health workshops have previously been shown to be effective in improving postpartum knowledge, performance of pelvic floor muscle exercises, and bowel-specific quality of life. Group learning through a class focused on behavioral modification and pelvic floor muscle exercises for women with urinary incontinence, has been shown to be an effective means to educate women about urinary incontinence management. The PAKS study hopes to demonstrate whether Spanish-speaking women that undergo an informative workshop on pelvic floor disorders via video in Spanish are more likely to raise their level of knowledge surrounding pelvic floor disorders and improve the pelvic floor symptoms.

DETAILED DESCRIPTION:
Purpose: The purpose of this study is to determine if an informational workshop on pelvic floor disorders administered via a video intervention will increase Spanish-speaking women's knowledge of pelvic floor disorders and decrease pelvic floor symptoms post-intervention.

Hypothesis or Aim: A single 20 minute video workshop on pelvic floor disorders will improve Spanish-speaking women's knowledge of pelvic floor disorders immediately post-intervention and at 4 weeks post-intervention compared to a pre-intervention knowledge.

Justification of the Study (Background): It is estimated that by the year 2050 in the United States, 58.2 million women will have at least 1 pelvic floor disorder. However, understanding of these disorders among patients is low. Prior studies assessing patient knowledge have shown that participants often did not understand basic urogynecologic terms such as urinary incontinence, pelvic organ prolapse, and pelvic floor disorder and that the participants had poor knowledge of participants' conditions.

Latinos will comprise 30% of the population in the United States by year 2060. In Hispanic women, barriers such as lower income, lower education, limited English language proficiency and lack of health coverage influence access to health care. In those with pelvic floor disorders, additional barriers such as poor understanding of general medical conditions, medical terminology, and female anatomy may lead to low understanding of participants' condition, treatment options, and therapies. Given this high prevalence estimate, educating and optimizing care for Hispanic women with such disorders is imperative with implications of having a significant societal impact.

Pelvic floor health workshops have previously been shown to be effective in improving postpartum knowledge, performance of pelvic floor muscle exercises, and bowel-specific quality of life. Learning through a class focused on behavioral modification and pelvic floor muscle exercises for women with urinary incontinence, was shown to be an effective means to educate women about urinary incontinence management. Women's knowledge, symptoms, and quality-of-life scores significantly improved at 3 months after undergoing an educational pelvic health workshop on incontinence and pelvic organ prolapse.

Currently, no studies have investigated the effects of a formal educational pelvic floor disorder workshop in Spanish on this knowledge or its impact on patient symptoms in those who suffer from pelvic floor disorders at baseline. The investigators research project proposes to close the gap between patient knowledge and scientific knowledge and potentially improve pelvic floor symptoms. The investigators' video workshop will empower women with knowledge and allow the women to make informed decisions surrounding the women's pelvic floor health. It will provide the women with tools to improve the women's own pelvic floor health. A pelvic floor health workshop targeted to Spanish-speaking women is an innovative concept which could lead to better patient care in a growing population. It may be the first step in prevention of future pelvic floor conditions.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years or older
* Interested in learning about pelvic floor disorders
* Spanish-speaking.

Exclusion Criteria:

* Women under 18 years of age
* Have previously completed the Prolapse and Incontinence Knowledge Questionnaire
* Unable to speak Spanish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 114 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Pelvic Floor Knowledge Scores Immediately Postintervention | Immediately after intervention administered
  Difference in questionnaire scores based on the validated Spanish version of the Prolapse and Incontinence Knowledge Questionnaire from baseline compared to immediately post-intervention after an educational video workshop.
  The Prolapse and Incontinence Knowledge Questionnaire is a 24-item condition-specific questionnaire that consists of 2 knowledge subscales: questions concerning pelvic organ prolapse (score range 0-12) and urinary incontinence (score range 0-12). Each item is given a score of 1 if answered correctly and 0 if answered incorrectly. Women are given a score of 0 if they answered "I don't know" or "No lo sé" presuming a lack of knowledge. Higher scores mean greater knowledge of these pelvic floor disorders.

SECONDARY OUTCOMES:
Pelvic Floor Knowledge Scores at 4 Weeks Postintervention | At 4 weeks postintervention
  Difference in questionnaire scores based on the validated Spanish version of the Prolapse and Incontinence Knowledge Questionnaire from baseline compared to 4 weeks post-intervention after an educational video workshop
  The Prolapse and Incontinence Knowledge Questionnaire is a 24-item condition-specific questionnaire that consists of 2 knowledge subscales: questions concerning pelvic organ prolapse (score range 0-12) and urinary incontinence (score range 0-12). Each item is given a score of 1 if answered correctly and 0 if answered incorrectly. Women are given a score of 0 if they answered "I don't know" or "No lo sé" presuming a lack of knowledge. Higher scores mean greater knowledge of these pelvic floor disorders.
Pelvic Floor Symptom Scores at 4 Weeks Postintervention | At 4 weeks postintervention
  Difference in Pelvic Floor Distress Inventory-20 questionnaire scores at 4 weeks postintervention from baseline compared to 4 weeks post-intervention after an educational video workshop
  The Pelvic Floor Distress Inventory-20 is a set of 20 symptom questions, answered on a 4-point Likert scale: 1 = not at all to 4 = quite a bit. The mean values of all answered items are multiplied by 25 to determine the scale score (range 0-100). A summary score is also reported (range 0-300). Higher scores denote a greater symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Keila S Muniz, MD, Study Director — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu JM, Hundley AF, Fulton RG, Myers ER. Forecasting the prevalence of pelvic floor disorders in U.S. Women: 2010 to 2050. Obstet Gynecol. 2009 Dec;114(6):1278-1283. doi: 10.1097/AOG.0b013e3181c2ce96. PMID 19935030
- [Background] Hawary A, Sinclair A, Pearce I. The origin of information: are IUGA-specific patient information leaflets the answer? Int Urogynecol J. 2010 Aug;21(8):1001-4. doi: 10.1007/s00192-010-1142-0. Epub 2010 Apr 17. PMID 20401466
- [Background] Senekjian L, Heintz K, Egger MJ, Nygaard I. Do Women Understand Urogynecologic Terminology? Female Pelvic Med Reconstr Surg. 2011 Sep;17(5):215-217. doi: 10.1097/SPV.0b013e31822dcffe. PMID 21984964
- [Background] Good MM, Korbly N, Kassis NC, Richardson ML, Book NM, Yip S, Saguan D, Gross C, Evans J, Harvie HS, Sung V; Society of Gynecologic Surgeons Fellows Pelvic Research Network. Prolapse-related knowledge and attitudes toward the uterus in women with pelvic organ prolapse symptoms. Am J Obstet Gynecol. 2013 Nov;209(5):481.e1-6. doi: 10.1016/j.ajog.2013.06.001. Epub 2013 Jun 5. PMID 23748108
- [Background] Colby SL, Ortman JM. Projections of the size and composition of the U.S. population: 2014 to 2060. Population Estimates 2015. https://www.census.gov/content/dam/Census/library/ publications/2015/demo/p25-1143.pdf. Accessed October 23, 2017.
- [Background] Roberts RE, Lee ES. Medical care use by Mexican-Americans: evidence from the human population laboratory studies. Med Care. 1980 Mar;18(3):267-81. PMID 7366256
- [Background] Andersen R, Lewis SZ, Giachello AL, Aday LA, Chiu G. Access to medical care among the Hispanic population of the southwestern United States. J Health Soc Behav. 1981 Mar;22(1):78-89. No abstract available. PMID 7240708
- [Background] Freeman G, Lethbridge-Cejku M. Access to health care among Hispanic or Latino women: United States, 2000-2002. Adv Data. 2006 Apr 20;(368):1-25. PMID 16646390
- [Background] Insaf TZ, Jurkowski JM, Alomar L. Sociocultural factors influencing delay in seeking routine health care among Latinas: a community-based participatory research study. Ethn Dis. 2010 Spring;20(2):148-54. PMID 20503895
- [Background] Khan AA, Sevilla C, Wieslander CK, Moran MB, Rashid R, Mittal B, Maliski SL, Rogers RG, Anger JT. Communication barriers among Spanish-speaking women with pelvic floor disorders: lost in translation? Female Pelvic Med Reconstr Surg. 2013 May-Jun;19(3):157-64. doi: 10.1097/SPV.0b013e318288ac1c. PMID 23611934
- [Background] Hyakutake MT, Han V, Baerg L, Koenig NA, Cundiff GW, Lee T, Geoffrion R. Pregnancy-Associated Pelvic Floor Health Knowledge and Reduction of Symptoms: The PREPARED Randomized Controlled Trial. J Obstet Gynaecol Can. 2018 Apr;40(4):418-425. doi: 10.1016/j.jogc.2017.10.022. PMID 29680079
- [Background] Gerard L. Group learning behavior modification and exercise for women with urinary incontinence. Urol Nurs. 1997 Mar;17(1):17-22. PMID 9110901
- [Background] Geoffrion R, Robert M, Ross S, van Heerden D, Neustaedter G, Tang S, Milne J. Evaluating patient learning after an educational program for women with incontinence and pelvic organ prolapse. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Oct;20(10):1243-52. doi: 10.1007/s00192-009-0919-5. Epub 2009 Jun 11. PMID 19517050
- [Background] Shah AD, Massagli MP, Kohli N, Rajan SS, Braaten KP, Hoyte L. A reliable, valid instrument to assess patient knowledge about urinary incontinence and pelvic organ prolapse. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Sep;19(9):1283-9. doi: 10.1007/s00192-008-0631-x. Epub 2008 May 15. PMID 18480958